CLINICAL TRIAL: NCT00927745
Title: Long Term Clinical Evaluation of AutoFlow Mode During Assist-Controlled Ventilation in ICU Patients
Brief Title: Clinical Evaluation of AutoFlow Mode During Mechanical Ventilation
Acronym: AFON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Victor Dupouy (Other)
Responsible Party: Maurice TOULLALAN, Director, Centre Hospitalier Victor Dupouy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AFON study
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Ventilation, Mechanical
Keywords: Respiration Artificial; Positive-Pressure Respiration; Critical Care; Intensive Care Units
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With AutoFlow (Experimental): Assist-controlled ventilation with activation of AutoFlow mode
  Interventions: Device: AutoFlow mode on Evita 4 Dräger ventilators
- Without AutoFlow (Active Comparator): Assist-controlled ventilation without activation of AutoFlow mode
  Interventions: Device: Evita 4 Dräger ventilators

INTERVENTIONS:
Device: AutoFlow mode on Evita 4 Dräger ventilators — Activation of AutoFlow mode during assist-controlled ventilation
  Arms: With AutoFlow
Device: Evita 4 Dräger ventilators — Assist-controlled ventilation without activation of AutoFlow mode
  Arms: Without AutoFlow

SUMMARY:
The purpose of this study is to evaluate the long term use of AutoFlow mode during mechanical ventilation in ICU patients

DETAILED DESCRIPTION:
Many new mechanical ventilation modes are proposed without clinical evaluation. Among them, "dual-controlled" modes, as AutoFlow, are supposed to improve patient-ventilator interfacing, and could led to lesser alarm. This study is a long term clinical evaluation of AutoFlow during assist-controlled ventilation, focusing on its efficacy (on gas exchange and outcome) and on ventilator alarms.

ELIGIBILITY:
Inclusion Criteria:

* adult patients under assist-controlled ventilation with an Evita 4 ventilator (Dräger, France) for an expected duration of more than two days

Exclusion Criteria:

* coma
* ventilation longer than 12 hours prior to inclusion
* pregnancy
* inclusion in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2002-12; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
gas exchange | daily during mechanical ventilation
sedation length | ICU discharge
ventilator alarm rates | daily during mechanical ventilation

SECONDARY OUTCOMES:
length of mechanical ventilation | ICU discharge
ventilator asssociated pneumonia rate | ICU discharge
SOFA score | daily during mechanical ventilation
death rate | ICU discharge
cumulative sedation drugs dosage | ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hervé MENTEC, MD, Study Director — Centre Hospitalier Victor Dupouy
Locations (1):
- Centre Hospitalier Victor Dupouy, Argenteuil, France